CLINICAL TRIAL: NCT05946616
Title: Probing Mechanisms of Procedural Memory Transformation With Cross-frequency Transcranial Alternating Current Stimulation (Cf-tACS) as an Avenue to Sculpt Sensorimotor Behavior
Brief Title: Spectral Characteristics of Memory Transformation
Acronym: MEM_MOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 00126392
Record Dates: First submitted 2023-06-30; First posted 2023-07-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Behavior Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active non-invasive brain stimulation during behavioral memory interference (Experimental): Non-invasive brain stimulation with transcranial alternating current stimulation will be applied during a memory interference intervention.
  Interventions: Other: Transcranial alternating current stimulation (tACS) combined with behavioral intervention
- Sham stimulation during behavioral memory interference (Sham Comparator): Inactive (sham) stimulation will be applied during a memory interference intervention.
  Interventions: Other: Inactive (sham) stimulation combined with behavioral intervention

INTERVENTIONS:
Other: Transcranial alternating current stimulation (tACS) combined with behavioral intervention — Transcranial alternating current stimulation (tACS) combined with behavioral intervention (memory interference).
  Arms: Active non-invasive brain stimulation during behavioral memory interference
Other: Inactive (sham) stimulation combined with behavioral intervention — Inactive (sham) stimulation combined with behavioral intervention (memory interference)
  Arms: Sham stimulation during behavioral memory interference

SUMMARY:
Sometimes, it is necessary to re-learn a previously learned movement behavior, for example, a bad posture during the golf drive or while playing the piano. Unlearning or relearning an intensively trained behavior is particularly important if the behavior is hampering recovery, for example, in chronic pain or after a stroke. With this pilot study, the brain mechanisms that control the change of pre-existing stable memories of a motor skill will be tested with electroencephalography (EEG). Non-invasive brain stimulation will be used to modulate these brain mechanisms and test if it is possible to change the pre-existing motor memory and the learning of a new motor skill.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (2/3 of the final sample will be ≥60years of age)
* No previous stroke, brain tumor, neurodegenerative disease, or trauma to the head
* Ability to give consent for study participation
* who have access to a personal computer with internet

Exclusion Criteria:

* • Pregnancy

  * Inability to use all ten fingers to type on a standard computer keyboard
  * Uncorrected vision, hindering perception of visual cues presented on a standard computer screen
  * Medication use at the time of study that may interfere with learning or the effect of tACS, including but not limited to carbamazepine, flunarizine, sulpiride, rivastigmine, dextromethorphan;
  * Neuromuscular disorders affecting hand and finger movements necessary for 10-finger keyboard typing
  * Presence of neurological or psychiatric disorders
  * Presence of scalp injury or disease
  * Prior history of seizures
  * Prior intracranial surgery
  * Prior brain radiotherapy
  * Prior history of intracranial tumor, intracranial infection, or cerebrovascular malformation
  * Metal in head or neck
  * Contraindications to MRI (such as severe claustrophobia, implanted medical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral: interference rate | before - after one single intervention (1 hour)
  Change in performance precision of a previously learned sensorimotor skill
Neural: brain connectivity change | before - after one single intervention (1 hour)
  Change in EEG-derived markers of brain activation and connectivity

SECONDARY OUTCOMES:
Behavioral: interference rate | before - after one single intervention (24 hour follow-up)
  Change in performance precision of a previously learned sensorimotor skill
Neural: brain connectivity change | before - after one single intervention (24 hour follow-up)
  Change in EEG-derived markers of brain activation and connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin-Friederike Heise, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States